CLINICAL TRIAL: NCT01873482
Title: Traditional African Healing Ceremony in a U.S. Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00042492
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Fatigue Syndrome; Anxiety; Depression; Cancer
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Anxiety Disorders; Depression; Neoplasms

ARMS (1):
- Movement with rhythm (Experimental): Subjects will move for 1 hour in time to the Congolese rhythm called Zebola.
  Interventions: Behavioral: Movement to rhythm

INTERVENTIONS:
Behavioral: Movement to rhythm — Movement to rhythm

SUMMARY:
Pre-agricultural societies almost universally used healing ceremonies that involved reverence, rhythm and dance in the presence of a healer. It is believed that we are "wired" for such experiences and they foster an integrative mode of consciousness similar to that of mindfulness based stress reduction, which has been shown to have therapeutic effects in a variety of conditions. Collaborator Ava Lavonne Vinesett of the Duke Dance Program has developed a healing ceremony based in sub-Saharan African traditions. The investigators plan is to have 25 subjects with a variety of clinical conditions participate in this ceremony. Subjects will then be asked to write a commentary about their experience and to participate in a focus group discussion. It is anticipated that the study will give us some idea of how promising this approach would be and what kinds of patients might benefit. Safety issues are minimal and include the possibility of injury (though the dancing is not strenuous) and psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 65 with one of the diagnoses listed above or with 8 visits to their provider in the last year and with no diagnosis of chronic illness.

Exclusion Criteria:

* physical disability making participation difficult and previous experience with a similar ceremony, for instance while growing up in Africa.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Report from each participant as to whether they found the experience positive, neutral or negative. | During the first hour after the intervention

SECONDARY OUTCOMES:
written narrative of experience | During the first hour after the intervention

OTHER OUTCOMES:
Encounter group discussion | During the first hour after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wilson, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States